CLINICAL TRIAL: NCT07228104
Title: Adjuvant STeRoid Outcomes in Idiopathic Subglottic Stenosis
Brief Title: Use of Steroid Injections to Prevent the Recurrence of Tracheal Stenosis in Idiopathic Subglottic Stenosis
Acronym: ASTRO
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00507375; 1UG3HL173394-01A1 (NIH)
Record Dates: First submitted 2025-11-11; First posted 2025-11-14 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Idiopathic Subglottic Stenosis
Keywords: Steroid injection; Stenosis
MeSH Terms: conditions — Idiopathic subglottic tracheal stenosis; Constriction, Pathologic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intralesional steroid injection with Triamcinolone (Experimental)
  Interventions: Drug: Triamcinolone 0.1%
- Intralesional Placebo injection (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Triamcinolone 0.1% — Intralesional Triamcinolone injection 3x at one, two, and three months following surgical dilation
  Arms: Intralesional steroid injection with Triamcinolone
Drug: Placebo — Intralesional Placebo injection 3x at one, two, and three months following surgical dilation
  Arms: Intralesional Placebo injection

SUMMARY:
This study will examine the ability of steroid injections into the site of stenosis following surgical dilation to delay the need for repeated surgical dilations.

ELIGIBILITY:
Inclusion Criteria:

* Have a life expectancy of ≥6 months; and,
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1.

Exclusion Criteria:

* History of subglottic stenosis from identifiable cause (not idiopathic), including any of the below clinical criteria:
* Prolonged endotracheal intubation or tracheostomy (intervention greater than 7 days immediately prior to diagnosis of subglottic stenosis);
* External physical trauma (including but not limited to blunt, penetration, chemical, or thermal injury) that causes injury to the subglottis;
* Clinical diagnosis of granulomatosis with polyangiitis (GPA);
* Radiation exposure to the neck;
* Current or previous treatment with Serial Intralesional Steroid Injection (SILSI);
* Use of systemic corticosteroids (oral, intravenous, or intramuscular glucocorticoids), regardless of indication, within 7 days before triamcinolone administration;
* Local administration of corticosteroids (ophthalmic, intranasal, inhaled) is not prohibited. However, the administration of intraarticular corticosteroids during the treatment phase is not recommended due to potential increased risk of infection.
* Intralesional administration, in a site other than the subglottis, of corticosteroids should be discussed with the site PI before enrollment
* Intraarticular corticosteroids during the treatment phase due to potential increased risk of infection;
* Use of anticoagulants other than aspirin (aspirin dose should not exceed 81mg);
* Pulmonary disease including interstitial lung disease and Chronic Obstructive Pulmonary Disease (COPD)/emphysema;
* Systemic infection requiring treatment with antibiotics, antifungal, or antiviral agents within 21 days of enrollment;
* Poorly controlled diabetes as defined by a HbA1C value greater or equal to 8.0 in the last 180 days);
* Participants with active cancer or a history of cancer in the last 5 years, except for squamous or basal cell carcinoma of the skin;
* Participation in any clinical trial involving an investigational drug or device, within four weeks, or 5 half-lives of the investigational agent (whichever time point is longer) prior to enrollment or during this trial participation;
* Active autoimmune disease requiring systemic treatment;
* History of solid organ transplant due to use of immunosuppression;
* Contraindication to any aspect of the index endoscopic dilation procedure.
* Inability to tolerate in office SILSI procedure;
* Contraindication, hypersensitivity, or history of intolerance to oral or injectable steroids;
* Contraindication to intralipid including:
* Severe lipid metabolism disorders characterized by hypertriglyceridemia;
* Hypersensitivity to eggs, soybean, peanut protein, or any active ingredient in intralipid;
* History of intolerance to intralipid;
* Participants with known, suspected, or plan for becoming pregnant or breastfeeding;
* New York Heart Association (NYHA) class II-IV heart failure within the past 6 months;
* History of angioedema;
* History of subglottic stenosis from other causes, including prolonged intubation (intubation of >1 week immediately prior to diagnosis of subglottic stenosis, external physical trauma that causes injury to the subglottis);
* Lack of capacity to consent;
* Alcohol or substance abuse or dependence in the past 6 months;
* Participants who for any reason may not complete the study as judged by the PI;
* Participants planning to move to another city or state during the duration of the study;
* Not able to undergo phlebotomy as reported by the participant or determined by the study coordinator or physician.
* The presence of a medical condition, and/or use of a medication and/or any substance, individually or in aggregate, that in the judgement of the study team could impair study participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2031-01-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Change in Peak Expiratory Flow (Liters/min) | 6 Months

SECONDARY OUTCOMES:
Clinical COPD Questionnaire | 6 months
  Score range 0-60, Lower score indicates better health
Voice Handicap Index-10 | 6 Months
  Score range 0 to 40, Lower score indicates better voice

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Hillel, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF